CLINICAL TRIAL: NCT06567535
Title: A Single-arm, Single-center Clinical Study of Endoscopic Combined With Intraoperative Navigation-assisted Treatment of Giant Mandibular Cysts
Brief Title: Treatment of Mandibular Bone Cyst by Navigation and Endoscopy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2024-261-03
Record Dates: First submitted 2024-07-11; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Jaw Cysts
MeSH Terms: conditions — Jaw Cysts | interventions — Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Navigation and endoscopy Group (Experimental): Preoperative copies of the patient's maxillofacial imaging data were digitally designed, professional software was used to segment cystic lesions and segment the inferior alveolar nerve together, and then the data was imported into the navigation system. The surgeon placed a mandibular reference frame in the anterior mandibular region, and used the navigation probe to accurately locate the difficult areas such as the anterior part of the capsule cavity, the apical part of the tooth root and the ascending branch of the mandible under the guidance of navigation. After accurate positioning was obtained, the navigation adapter was loaded onto the endoscope to locate the lesions in all directions and the inferior alveolar nerve under visual conditions, and further precisely curettage the lesions in the cystic cavity with the assistance of the adapter.
  Interventions: Procedure: Navigation and endoscopy

INTERVENTIONS:
Procedure: Navigation and endoscopy — The model was reconstructed using patient CT data, and intraoperative surgery was performed using endoscopy and navigation.

SUMMARY:
In this study, with the assistance of endoscopic technology and intraoperative navigation technology, the removal and curettage of large odontogenic jaw cyst occurred in the mandible were performed to reduce the rate of postoperative nerve injury. In this study, the investigators compared the efficacy of traditional extraction and curettage with endoscopic navigation assistance in the treatment of giant mandibular bone cysts. In this study, the rate of inferior alveolar nerve injury 1 month after surgery was taken as the main outcome index, and the recurrence rate 1 year after surgery was taken as the secondary outcome index, to explore whether endoscopic combined with intraoperative navigation-assisted treatment of giant mandibular bone cyst could achieve lower postoperative nerve injury rate and postoperative recurrence rate.

DETAILED DESCRIPTION:
This study hypothesized that endoscopy combined with intraoperative navigation-assisted treatment of giant mandibular bone cysts was more effective than the traditional surgical method of removal and curettage. In this study, a prospective, single-arm, Phase II clinical study was used to design the protocol, and the estimated rate of postoperative nerve injury was reduced by about 12% from 32% to 20% compared with traditional surgery. This study started from the recruitment of subjects, oral panoramic film, maxillofacial CT and other imaging examinations were performed to confirm the diagnosis. After preliminary screening according to the inclusion and exclusion criteria, patients were enrolled after signing the informed consent letter. Endoscopic and navigational techniques were used for surgical treatment. This study referred to the prospective study of Abdullah Hanfesh et al. to evaluate the function of the inferior alveolar nerve: the bilateral mandibular and lower lip were divided into four areas: area A, area B, area C, and area D. The four areas will be lightly touched, acupuncture, cold and hot stimulation, and two-point discrimination detection four times respectively, and the detection situation of each area will be recorded. Inferior alveolar nerve function was detected before and 1 month after surgery. Light touch detection 4 points, acupuncture detection 1 point, hot and cold stimulation 1 point, two-point discrimination detection 5 points showed no nerve damage. Any other score for any of the above is considered to be nerve damage. The main study measure: postoperative nerve injury rate was calculated until the last subject was followed up. The main efficacy index of this study was the postoperative nerve injury rate of endoscopic combined with intraoperative navigation-assisted treatment of giant mandibular bone cysts. The hypothesis of this study is that the postoperative nerve injury rate of endoscopy combined with intraoperative navigation-assisted treatment of giant mandibular cyst is lower than that of traditional excision and curettage. Study parameters were set as follows: α=0.025 (unilateral) and Power=80%. According to the results of previous studies or pre-tests, the postoperative nerve injury rate of the endoscopic navigation group was reduced by about 20% to 12%. 109 cases were calculated using PASS 15.0 software, and 122 subjects were included considering the 10% shedding rate.

ELIGIBILITY:
Inclusion Criteria:

1. They are between 18 and 75 years old
2. Imaging and puncture pathology showed odontogenic cystic lesion of the mandible
3. Cystic lesions greater than or equal to 2cm in diameter and spread to the inferior alveolar nerve
4. New or recurrent cyst lesions, or odontogenic cystic lesions that are still greater than or equal to 2cm after other treatment such as fenestration and affecting the lower alveolar nerve
5. No serious systemic disease, tolerant of general anesthesia
6. Patients undergoing surgical treatment for mandibular bone cysts under general anesthesia
7. There was no inferior alveolar nerve injury before operation
8. Have not participated in other clinical trials within 30 days
9. Patients who volunteer to participate in the program and sign informed consent

Exclusion Criteria:

1. The patient has severe systemic disease or pregnancy, and is judged to be unable to tolerate the course of this clinical study and cannot tolerate general anesthesia after evaluation by the research team and multidisciplinary consultation
2. Inability to complete the entire clinical research process due to personal, social, and economic reasons
3. Patients with psychiatric disorders or inability to perceive and communicate normally, such as schizophrenia, claustrophobia, etc., are unable to complete the examination and cooperate in the entire clinical research process

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2024-08-20 (Estimated); Primary Completion 2026-11-10 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Rate of inferior alveolar nerve injury at one month postoperatively | one month
  Rate of inferior alveolar nerve injury at one month postoperatively

SECONDARY OUTCOMES:
Recurrence rate one year after surgery | one year
  Recurrence rate one year after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Yan Wang, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- WangYan, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rajendra Santosh AB. Odontogenic Cysts. Dent Clin North Am. 2020 Jan;64(1):105-119. doi: 10.1016/j.cden.2019.08.002. Epub 2019 Oct 18. PMID 31735221
- [Result] Manor E, Kachko L, Puterman MB, Szabo G, Bodner L. Cystic lesions of the jaws - a clinicopathological study of 322 cases and review of the literature. Int J Med Sci. 2012;9(1):20-6. doi: 10.7150/ijms.9.20. Epub 2011 Nov 9. PMID 22211085
- [Result] Anavi Y, Gal G, Miron H, Calderon S, Allon DM. Decompression of odontogenic cystic lesions: clinical long-term study of 73 cases. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2011 Aug;112(2):164-9. doi: 10.1016/j.tripleo.2010.09.069. Epub 2010 Dec 30. PMID 21194990
- [Result] Marin S, Kirnbauer B, Rugani P, Mellacher A, Payer M, Jakse N. The effectiveness of decompression as initial treatment for jaw cysts: A 10-year retrospective study. Med Oral Patol Oral Cir Bucal. 2019 Jan 1;24(1):e47-e52. doi: 10.4317/medoral.22526. PMID 30573706
- [Result] Wang Y, Chang S, Lin Z, Chen R, Huang Z. Endoscopic-assisted enucleation of large mandibular odontogenic cysts. Oral Surg Oral Med Oral Pathol Oral Radiol. 2020 Feb;129(2):115-119. doi: 10.1016/j.oooo.2019.05.012. Epub 2019 Jun 6. PMID 31786170
- [Result] Tamiolakis P, Thermos G, Tosios KI, Sklavounou-Andrikopoulou A. Demographic and Clinical Characteristics of 5294 Jaw Cysts: A Retrospective Study of 38 Years. Head Neck Pathol. 2019 Dec;13(4):587-596. doi: 10.1007/s12105-019-01011-7. Epub 2019 Feb 13. PMID 30758760
- [Result] Wakolbinger R, Beck-Mannagetta J. Long-term results after treatment of extensive odontogenic cysts of the jaws: a review. Clin Oral Investig. 2016 Jan;20(1):15-22. doi: 10.1007/s00784-015-1552-y. Epub 2015 Aug 8. PMID 26250795
- [Result] Gao Z, Ni QW, Gao W, Liu YP, Zhang Q. Application of endoscopy to treat mandibular keratocystic odontogenic tumors. Braz J Med Biol Res. 2017 Jul 10;50(8):e6209. doi: 10.1590/1414-431X20176209. PMID 28700034
- [Result] Sembronio S, Albiero AM, Zerman N, Costa F, Politi M. Endoscopically assisted enucleation and curettage of large mandibular odontogenic keratocyst. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2009 Feb;107(2):193-6. doi: 10.1016/j.tripleo.2008.07.020. Epub 2008 Sep 17. PMID 18801672
- [Result] Huang Z, Huang Z, Zhang D, Hu H, Liang Q, Chen W. Endoscopically-assisted operations in the treatment of odontogenic peripheral osteomyelitis of the posterior mandible. Br J Oral Maxillofac Surg. 2016 Jun;54(5):542-6. doi: 10.1016/j.bjoms.2016.02.023. Epub 2016 Mar 26. PMID 27025231
- [Result] Azarmehr I, Stokbro K, Bell RB, Thygesen T. Surgical Navigation: A Systematic Review of Indications, Treatments, and Outcomes in Oral and Maxillofacial Surgery. J Oral Maxillofac Surg. 2017 Sep;75(9):1987-2005. doi: 10.1016/j.joms.2017.01.004. Epub 2017 Jan 18. PMID 28193444
- [Result] Sukegawa S, Kanno T, Furuki Y. Application of computer-assisted navigation systems in oral and maxillofacial surgery. Jpn Dent Sci Rev. 2018 Aug;54(3):139-149. doi: 10.1016/j.jdsr.2018.03.005. Epub 2018 May 7. PMID 30128061
- [Result] de Geer AF, Brouwer de Koning SG, van Alphen MJA, van der Mierden S, Zuur CL, van Leeuwen FWB, Loeve AJ, van Veen RLP, Karakullukcu MB. Registration methods for surgical navigation of the mandible: a systematic review. Int J Oral Maxillofac Surg. 2022 Oct;51(10):1318-1329. doi: 10.1016/j.ijom.2022.01.017. Epub 2022 Feb 11. PMID 35165005
- [Result] Sozzi D, Filippi A, Canzi G, De Ponti E, Bozzetti A, Novelli G. Surgical Navigation in Mandibular Reconstruction: Accuracy Evaluation of an Innovative Protocol. J Clin Med. 2022 Apr 6;11(7):2060. doi: 10.3390/jcm11072060. PMID 35407667
- [Result] Hanfesh A, Salma RG, Al Mutairi K, AlShiha SK, Al Otaibi S. The neurosensory deficit of inferior alveolar nerve following bilateral sagittal split osteotomy: a prospective study. Oral Maxillofac Surg. 2022 Sep;26(3):401-415. doi: 10.1007/s10006-021-01005-2. Epub 2021 Sep 12. PMID 34510239

DOCUMENTS (1):
  • Study Protocol (2024-05-25): https://cdn.clinicaltrials.gov/large-docs/35/NCT06567535/Prot_000.pdf